CLINICAL TRIAL: NCT05507632
Title: A Prospective, Single-arm, Phase II Clinical Study of the Efficacy and Safety of Donafenib Plus Sintilimab Combined With Transarterial Chemoembolization (TACE) in Patients With BCLC Stage B/C Hepatocellular Carcinoma
Brief Title: Donafenib Plus Sintilimab in Combination With TACE in Patients With Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-256
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; HCC; Donafenib; Sintilimab; transarterial chemoembolisation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Experimental): All patients treatment with Donafenib plus Sintilimab in combination with TACE
  Interventions: Combination Product: Donafenib plus Sintilimab in combination with transarterial chemoembolisation

INTERVENTIONS:
Combination Product: Donafenib plus Sintilimab in combination with transarterial chemoembolisation — Donafenib plus Sintilimab in combination with transarterial chemoembolisation (TACE)

SUMMARY:
To evaluate the efficacy and safety of Donafenib plus Sintilimab in combination with transarterial chemoembolisation (TACE) in patients with unresectable hepatocellular carcinoma(HCC).

DETAILED DESCRIPTION:
Transarterial chemoembolisation (TACE) was effective and safe for hepatocellular carcinoma. Donafenib was better than sorafenib in overall survival in untreated advanced hepatocellular carcinoma, and programmed cell death protein-1 (PD-1) antibody was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has evaluated TACE plus donafenib and sintilimab. Thus, the investigators carried out this prospective, single-arm study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily joins the study and signs an informed consent;
* Aged 18 to 75 years, both men and women;
* Clinical diagnosis of BCLC B(4 <=tumor numbers<=10 ) or C-stage hepatocellular carcinoma, no further first-line treatment;
* At least one intrahepatic evaluable tumor existed, intrahepatic tumor is the primary tumor burden;
* Child-Pugh score small or equal to 7 points (Child-Pugh A-B);
* The maximum liver tumor diameter < 7cm, All lesions in the liver could be treated with stage 1 or 2 TACE;
* Must be able to swallow tablets;
* ECOG score: 0 to 1 (according to the ECOG score classification);
* The expected survival is longer than 12 weeks;
* The laboratory parameters meets the following requirements (no blood components and cell growth factors are allowed within 14 days before the first dose):Absolute neutrophil count >= 1.5 x 10^9 / L; Platelets >= 50 x 10^9 / L; Hemoglobin >= 80 g / L; serum albumin >= 28 g / L; Thyroid stimulating hormone (TSH) <= 1 x ULN (if abnormalities should be considered at the same time FT3, FT4 levels, patients with FT3 and FT4 levels in normal range can also be enrolled); bilirubin <= 1.5 x ULN (within 7 days prior to the first dose); ALT <= 3 x ULN and AST <= 3 x ULN (within 7 days prior to the first dose); AKP <= 2.5 x ULN; serum creatinine <= 1.5 x ULN;
* For female that non-surgical sterilization or in childbearing age need to use a medically approved contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period; For female that non-surgical sterilization or in childbearing age must have a negative serum or urine HCG test within 72 hours prior to study enrollment; and must be non-lactating; for male patients whose partner in a childbearing age, effective methods of contraception should be given during the trial and at the end of Sintilimab injection.

Exclusion Criteria:

* The maximum liver tumor diameter >= 10 cm, tumor numbers > 10;
* Receive local treatment for HCC((e.g.,TACE, TAE, HAIC or radiotherapy); If the treatment of ablation and/or resection > 4 weeks is permitted;
* The patient has any active auto-immune disease or a history of auto-radioimmune disease; Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy;
* The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose > 10 mg/day of prednisone or other therapeutic hormones) and continues to be used within 2 weeks prior to enrollment;
* Known or suspected allergy to the investigational agents or any agent given in association with this trial;
* Known central nervous system tumors including metastatic brain disease;
* History of organ allograft;
* Ascites with clinical symptoms;
* The intrahepatic neoplasms showed diffuse changes;
* Suffering from hypertension, and cannot be well controlled by antihypertensive drugs (systolic blood pressure >= 140mmHg or diastolic blood pressure >=90 mmHg);
* Suffering heart diseases with clinical symptoms or those not well controlled, such as:(1) Heart failure in NYHA class 2 or higher;(2) Unstable angina;(3) Myocardial infarction occurred within 1 year;(4) Clinically symptomatic supraventricular or ventricular arrhythmia requiring treatment or intervention;(5) Tc > 450ms (male); QTc > 470ms (female).
* Abnormal coagulation (INR>2.0, PT extension time >4s), bleeding tendency or being treated with thrombolytic or anticoagulant therapy, allowing prophylactic use of low-dose aspirin and low-molecular-weight heparin;
* Evidence of bleeding diathesis; Patients with clinically significant gastrointestinal bleeding within 3 months prior to study entry.
* Events of arterial/venous thrombosis occurring within the first 6 months of enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Known history of hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliacs, coagulopathy, thrombocytopenia, etc.);
* Had intestinal obstruction and/or had clinical signs or symptoms of GI obstruction within 6 months prior to the start of study treatment, including incomplete obstruction related to pre-existing conditions or requiring routine parenteral hydration, parenteral nutrition, or tube feeding;
* Urine routine indicates that urine protein >= ++ and 24-hour urine protein amount > 1.0g was confirmed;
* The patient has active infection, unexplained fever (>=38.5 degree C) within 3 days before administration, or baseline white blood cell count > 15 x 10^9/L;
* Patients with congenital or acquired immunodeficiency (such as HIV-infected patients);
* HBV-DNA > 2000 IU/ml (or 10^4 copies/ml); or HCV-RNA > 10^3 copies/ml; or HBsAg+ and anti-HCV antibody positive patients;
* The patient has had other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
* Palliative radiotherapy for non-target lesions to control symptoms is permitted and must be completed at least 2 weeks prior to the start of the study treatment. The adverse events caused by radiotherapy have not recovered to <= CTCAE 1;
* Patients have previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or have received apatinib before;
* Inoculation of a live vaccine within less than 4 weeks prior to study or possibly during the study period;
* Pregnant or lactating women, or women of childbearing age who are unwilling to take contraceptive measures;
* According to the investigators, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory tests, abnormalities, accompanied by factors such as family or society, which may affect the safety of enrolled patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1

SECONDARY OUTCOMES:
The disease control rate (DCR) Duration of response DuraDuration of responsetion of response Duration of response | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1
Disease control rate (DOR) | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1
Progression free survival rate | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
  The progression free survival time defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1
Overall survival rate | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
  Overall survival rate is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes early.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhang Chen, Study Director — Nanfang Hostipal of Southern Medical University